CLINICAL TRIAL: NCT01377779
Title: Intercoat (Oxiplex/AP Gel) for Preventing Intrauterine Adhesions Following Operative Hysteroscopy for Suspected Retained Products of Conception - a Prospective Randomized Pilot Study
Brief Title: Efficiency of Intercoat (Oxiplex/AP Gel)in Decreasing Intrauterine Adhesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Moty Pansky, MD, Asaf Harofe MC
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2*13/09
Record Dates: First submitted 2011-06-15; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2009-07

CONDITIONS: Asherman Syndrome
Keywords: Oxiplex/AP gel; Prevention of Asherman's syndrome; Intra uterine adhesions
MeSH Terms: conditions — Gynatresia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intercoat treatment (Experimental): women treated by Intercoat gel following hysteroscopy for retained products of conception
  Interventions: Drug: Oxiplex/AP gel
- Control group (Placebo Comparator): No additional treatment following hysteroscopy was performed
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Oxiplex/AP gel — Intrauterine application of Intercoat following hysteroscopy
  Other Names: Intercoat
  Arms: Intercoat treatment
Drug: Normal Saline — No intrauterine application of Intercoat following hysteroscopy
  Other Names: Distention media
  Arms: Control group

SUMMARY:
This is a prospective single blind randomized controlled pilot study was designed to investigate whether the biological barrier Intercoat (Oxiplex/AP gel) reduces formation of intrauterine adhesions following hysteroscopic treatment for retained products of conception.

DETAILED DESCRIPTION:
Thirty women randomly divided equally into those who received Intercoat following hysteroscopic treatment for retained products of conception (study group) and those who did not receive the gel (controls). Safety and efficacy of the preparation were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Availability of the results of vaginal ultrasound or diagnostic hysteroscopy

Exclusion Criteria:

* Signs of infection upon admission
* Ongoing pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
safety of intrauterine application of Intercoat | 18 months
  women treated by Intercoat following their hysteroscopic procedure were followed for immediate and late adverse effects; fever, increased intrauterine adhesion formation upon follow up and changes in menstrual pattern

SECONDARY OUTCOMES:
efficacy of intrauterine application of Intercoat gel in reducing adhesion formation following hysteroscopic treatment for retained products of conception | 14 months
  intrauterine adhesions were graded according to the AFS score upon hysteroscopic follow up 6-8 weeks following initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Moty Pansky, MD, Principal Investigator — Asaf Harofe MC
Locations (1):
- Asaf Harofe MC, Ẕerifin, Israel